CLINICAL TRIAL: NCT07265908
Title: Establishment of a Biobank Aimed at Studying Gynecological Pathologies, of Male and Female Infertility and Pregnancy Pathologies
Brief Title: Biobank Aimed to Study Gynecological Pathologies, of Male and Female Infertility and Pregnancy Pathologies
Status: Enrolling by invitation | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Enrico Papaleo, Principal Investigator, IRCCS San Raffaele
Other Study IDs: REPRO-Biobank
Record Dates: First submitted 2025-09-17; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Gynecological Disorders; Male Infertility; Female Infertility; Pregnancy
MeSH Terms: conditions — Genital Diseases, Female; Infertility, Male; Infertility, Female | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The study involves the collection of surplus material in accordance with procedures within routine clinical practice, as well as the performance of additional procedures (blood sampling).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Affected participants: Subjects diagnosed with gynecological disorders, male or female infertility, or pregnancy-associated conditions.
  Interventions: Other: Blood sampling
- Healthy participants: Subjects without a diagnosis of gynecological disorders, male or female infertility, or pregnancy-associated conditions.
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Blood sampling

SUMMARY:
The REPRO-Biobank has been established at San Raffaele Hospital in Milan for the purpose of collecting and preserving human biological samples and associated data. Its primary objective is to support biomedical research, with a particular focus on advancing scientific knowledge - including in the field of genetics - related to gynecological disorders, male and female infertility, and pregnancy-related conditions.

ELIGIBILITY:
1. Affected participants

   Inclusion Criteria for adult patients (including pregnant and breastfeeding women) and pediatric patients affected by:
   * Male infertility
   * Female infertility
   * Gynecological disorders
   * Pregnancy-related conditions
   * Conditions requiring fertility preservation treatment (oocyte cryopreservation, ovarian tissue preservation)
   * Informed consent signed by the adult patient or by the parents/legal guardians of pediatric patients

   Exclusion Criteria
   * Patients unable or unwilling to sign the informed consent
2. Healthy participants Inclusion Criteria

   * Healthy adult subjects (including pregnant and lactating women)
   * Able to give informed consent for participation in the study

Exclusion Criteria

* Patients unable or unwilling to sign the informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: REPRO-Biobank anticipates the enrollment of approximately 300 individuals annually, comprising adult and pediatric patients diagnosed with gynecological disorders, male or female infertility, or pregnancy-related conditions, currently under care at the Gynecology and Obstetrics Unit / Centro Scienze della Natalità of San Raffaele Hospital, as well as healthy volunteers associated with the same Unit.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2043-12-31 (Estimated); Study Completion 2043-12-31 (Estimated)

PRIMARY OUTCOMES:
Developing a biobank/repository | Through study completion, an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Papaleo, MD, Principal Investigator — IRCCS San Raffaele
Locations (1):
- Irccs San Raffaele Hospital, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No